CLINICAL TRIAL: NCT01947387
Title: A Retrospective, Multi-Center Study Evaluating the Outcomes for Integra® Skin Sheet Bilayer or Single Layer Products Used in Complex Lower Extremity Soft Tissue Reconstruction
Brief Title: Retrospective Study Evaluating Outcomes for Integra® Skin Sheet Products in Lower Extremity Complex Wounds
Status: Completed | Type: Observational
Sponsor: Integra LifeSciences Corporation (Industry)
Collaborators: Georgetown University (Other)
Responsible Party: Sponsor
Other Study IDs: Integra 11-2011
Record Dates: First submitted 2013-08-12; First posted 2013-09-20 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-12

CONDITIONS: Complex Lower Extremity Soft Tissue Reconstruction

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (9):
- Integra
- Integra + NPWT (short-inpatient use only)
- Integra + NPWT (long-all other durations)
- Integra + STSG
- Integra + Dermoinductive Agent
- Free Flap
- Local Tissue Flap
- NPWT
- NPWT then Integra (on same admission)

SUMMARY:
This is a retrospective, multi-center study evaluating the outcomes of using Integra® skin sheet bilayer or single layer products for complex soft tissue reconstruction of lower extremity diabetic wounds compared to other treatments. Participating sites will collect information for all patients who received Integra, free flap, local tissue flap, or negative pressure therapy over a 5 year period. The patient must be a minimum of 1 year from index procedure, with index procedure being defined as the application of Integra, free flap, local tissue flap, or negative pressure. Any follow-up occurring during the year is eligible for inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic (I or II) male or female, age greater than 18 years
* Lower extremity wounds that required operative application of Integra, free flap, local tissue flap, or negative pressure wound therapy. Complex wounds are defined as wounds that involve exposed deep tissue (e.g. bone, tendon, fascia, ligament)
* The patient must be a minimum of 1 year from the index procedure, any follow-up occurring during the year is eligible for inclusion.

Exclusion Criteria:

* Age less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who received Integra, free flap, local tissue flap, or negative pressure wound therapy over a 5-year period. The patient must be a minimum of 1 year from the index procedure, any follow-up occurring during the year is eligible for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2013-08; Primary Completion 2014-09 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Wound recurrence rates after Integra application (and final split-thickness skin graft or dermoinductive agent application) as compared with free flap, local tissue flap, and negative pressure wound therapy. | 5 year period
  A dermoinductive agent is a product that is said to promote rapid wound healing.

SECONDARY OUTCOMES:
Time to ambulation/return to function after Integra application, free flap, local tissue flap, or negative pressure wound therapy. | 5 year period

OTHER OUTCOMES:
Time to wound bed preparation for receipt of a split thickness skin graft (STSG) or dermoinductive agent after having received Integra or negative pressure wound therapy | 5 years
Time to complete re-epithelization (as deemed by the surgeon) after Integra application or NPWT | 5 years

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Georgetown University Hospital Wound Healing Center, Washington D.C., District of Columbia
  - Northwestern University Feinberg School of Medicine Division of Plastic Surgery, Chicago, Illinois
  - Brigham and Women's Hospital, Inc, Boston, Massachusetts
  - University of Texas Southwestern Medical Ceter, Dallas, Texas